CLINICAL TRIAL: NCT01221090
Title: Employing Diabetes Self-Management Models to Reduce Health Disparities in Texas
Brief Title: Diabetes Self-Management Models to Reduce Health Disparities
Acronym: P20-P2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scott and White Hospital & Clinic (Other)
Collaborators: Texas A&M University (Other)
Responsible Party: Principal Investigator, Sam Forjuoh, Professor & Director of Research, Scott and White Hospital & Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 071304; P20MD002295 (NIH)
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Health disparities; Central Texas; PDA; CDSMP
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Personal Digital Assistant (Experimental): Individuals in this arm were taught to use a diabetes self-care software, Diabetes Pilot™ (Digital Altitudes, Arlington Heights, IL), developed for PalmOS® (Palm, Sunnyvale, CA) which was loaded on to compatible PDAs, the Tungsten™ E2 handheld device. The Diabetes Pilot allowed participants to monitor their blood glucose, blood pressure, medication usage, physical activity, and dietary intake by tracking these measures in an electronic diary.
  Interventions: Behavioral: PDA
- CDSMP (Active Comparator): 6-week, classroom-based program for diabetes self-management. The CDSMP, developed by Stanford University, equipped participants with the education and skill sets needed to take a more proactive approach in managing their chronic condition(s) and related symptoms.
  Interventions: Behavioral: CDSMP
- PDA/CDSMP (Active Comparator): Combined intervention
  Interventions: Behavioral: PDA/CDSMP
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: PDA — Technological assistance
  Other Names: Personal digital assistant
  Arms: Personal Digital Assistant
Behavioral: CDSMP — 6-week classes
  Other Names: Chronic disease self-management program
  Arms: CDSMP
Behavioral: PDA/CDSMP — Combined technology and education
  Other Names: PDA + CDSMP
  Arms: PDA/CDSMP

SUMMARY:
To evaluate the effectiveness of two different diabetes self-management approaches (Personal Digital Assistant-based intervention & Chronic Disease Self-Management Program) to reduce health disparities in minority, rural residents, and other underserved populations with type 2 diabetes in Central Texas. We hypothesise that: 1) Racial/ethnic minority patients with T2DM will be found to experience disparities in diabetes self-management treatment protocols and clinical outcomes, which persist even when controlling for age, gender, obesity, and insurance status; 2) Patients with T2DM who reside in more rural areas will be found to experience disparities in diabetes self-management treatment protocols and clinical outcomes as compared to more urban counterparts, controlling for age, gender, race/ethnicity, obesity, and insurance status; 3) The introduction of CSDMP and HIT protocols will improve diabetes-related self management behaviors, reduce HBA1c values, and increase quality of life in persons with T2DM as compared to controls. A combined intervention approach will result in the greatest reductions; 4) Health improvements following the introduction of CDSMP, HIT or CDSMP/HIT protocols in persons with T2DM compared to controls will be more marked in racial/ethnic minority patients and those patients residing in rural areas; 5) The introduction of self-management interventions will be cost-effective in reducing HbA1c values over time, and associated health care utilization including overall reduction in ER and acute care hospital admissions; 6) Although there is little prior research in this area to guide specific hypotheses, we hypothesize that, overall, there will be no significant cost-effective differential in CDSMP as compared to HIT approaches, although the cost-effective ratio may be stronger in particular subpopulations. The combined approach will have higher costs, but is also anticipated to have a higher cost-benefit ratio for minority populations; 7) The majority of clinicians will be willing to let their patients enroll in the study and will reinforce intervention protocols; and 8) These interventions can be embedded into existing health care structures. At the end of the study, Scott and White will institutionalize cost-effective treatment protocols.

DETAILED DESCRIPTION:
Despite concerted federal and state attempts to reduce health disparities over the past decades substantial disparities in reported rates of chronic disease for minorities still exist. In particular, African Americans and Hispanics experience higher rates of Type 2 diabetes (T2DM), and cardiovascular disease (CVD) than do other segments of the U.S. population. The objectives of this proposed research project are to test two different diabetes self-management (DSM) programs in a large multi-site health care organization in Central Texas that serves large populations of minority and rural residents, comparing outcomes in order to evaluate their efficacy for reducing health disparities. Our specific aims are to: 1) document the nature and magnitude of extant health disparities in diabetes treatment processes and outcomes; 2) evaluate different DSM intervention approaches on behavioral and clinical outcomes, with attention to differential effects by patient and environmental characteristics; 3) examine the cost-effectiveness of these different approaches to DSM education in minority and rural populations; and 4) explore the reach of our intervention efforts and the broader organizational impacts of DSM education, including feedback loops to clinicians and organizational receptivity to self-management approaches. Our study will employ four different activities: 1) an initial electronic chart review of 1300 records of adults; 2) a 2 by 2 open 24 month randomized clinical trial of behaviorally and technologically based DSM interventions with 400 adults age 21 and older who have type 2 diabetes (T2DM); 3) a cost-effectiveness analysis of the different treatment approaches; and 4) surveys of primary care providers and health care administrators. While our primary outcome will be reductions in hemoglobin A1c (HbA1c), our conceptual model includes clinical, behavioral, economic and organizational outcomes. We will also assess the extent to which our interventions reduce health disparities by examining differential treatment success. This study is innovative in its comparison of both behavioral and technological intervention approaches, its attention to the public health impact and cost-effectiveness of different intervention approaches, and its concern with organizational responses to intervention sustainability. A noteworthy significance will be the strengthening of the linkages between clinical and community treatment approaches and the identification of successful treatment strategies in different settings and populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM, including those who require insulin therapy, aged >18 years (eliminates the need to obtain assent for minors who are also dependent on their parents).
* Last measured HbA1c value of > 7.5% (this study hopes to show an improvement in the control of patient's diabetes, and not focused on patients who already show evidence of good disease control).
* Willingness and ability to attend one initial research visit and semi-annual routine follow-up visits over a 24-month period. The follow-up visits include height, weight, and blood pressure measurement and a survey. Surveys may be conducted by phone interview or mail when a follow-up visit can not be scheduled.
* Ability to read, write, and speak English at least at a grade 8 level so as to be able to engage in self-monitoring and use the commercial diabetes management software program (Diabetes Pilot), which is available only in English. For those with lower-literacy, assistance in filling out forms and understanding required intervention protocols will be provided, and use of a "buddy" will be recommended.

Exclusion Criteria:

* Not willing to sign an informed consent or be randomized to any of the four treatment/control groups, (we want to minimize any upfront treatment biases, while adhering to human subject protocols).
* Currently, documented severe alcoholism or drug abuse that is < 6 months ago (concerns that this problem is likely to significantly affect their ability and likelihood to comply with the study requirements over the course of the 24 months).
* Female patients who are pregnant or planning to become pregnant within 12 months (in pregnancy, type 2 diabetes is managed in a completely different manner than in non-pregnant patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel N Forjuoh, MD MPH DrPH, Principal Investigator — Scott & White
Locations (1):
- Scott & White Clinic, Temple, Texas, United States

REFERENCES:
- [Background] Vuong AM, Huber JC Jr, Bolin JN, Ory MG, Moudouni DM, Helduser J, Begaye D, Bonner TJ, Forjuoh SN. Factors affecting acceptability and usability of technological approaches to diabetes self-management: a case study. Diabetes Technol Ther. 2012 Dec;14(12):1178-82. doi: 10.1089/dia.2012.0139. Epub 2012 Sep 26. PMID 23013155
- [Background] Appiah B, Hong Y, Ory MG, Helduser JW, Begaye D, Bolin JN, Forjuoh SN. Challenges and opportunities for implementing diabetes self-management guidelines. J Am Board Fam Med. 2013 Jan-Feb;26(1):90-2. doi: 10.3122/jabfm.2013.01.120177. PMID 23288286
- [Result] Forjuoh SN, Huber C, Bolin JN, Patil SP, Gupta M, Helduser JW, Holleman S, Ory MG. Provision of counseling on diabetes self-management: are there any age disparities? Patient Educ Couns. 2011 Nov;85(2):133-9. doi: 10.1016/j.pec.2010.08.004. Epub 2010 Sep 21. PMID 20863646
- [Result] Forjuoh SN, Bolin JN, Gupta M, Huber C, Helduser JW, Holleman S, Robertson A, Ory MG. Disparities in diabetes management by race or ethnicity in a primary care clinic in central Texas. Tex Med. 2010 Nov 1;106(11):e1. PMID 21104573
- [Derived] Adepoju OE, Bolin JN, Phillips CD, Zhao H, Ohsfeldt RL, McMaughan DK, Helduser JW, Forjuoh SN. Effects of diabetes self-management programs on time-to-hospitalization among patients with type 2 diabetes: a survival analysis model. Patient Educ Couns. 2014 Apr;95(1):111-7. doi: 10.1016/j.pec.2014.01.001. Epub 2014 Jan 13. PMID 24468198
- [Derived] Forjuoh SN, Bolin JN, Huber JC Jr, Vuong AM, Adepoju OE, Helduser JW, Begaye DS, Robertson A, Moudouni DM, Bonner TJ, McLeroy KR, Ory MG. Behavioral and technological interventions targeting glycemic control in a racially/ethnically diverse population: a randomized controlled trial. BMC Public Health. 2014 Jan 23;14:71. doi: 10.1186/1471-2458-14-71. PMID 24450992
- [Derived] Adepoju OE, Bolin JN, Ohsfeldt RL, Phillips CD, Zhao H, Ory MG, Forjuoh SN. Can chronic disease management programs for patients with type 2 diabetes reduce productivity-related indirect costs of the disease? Evidence from a randomized controlled trial. Popul Health Manag. 2014 Apr;17(2):112-20. doi: 10.1089/pop.2013.0029. Epub 2013 Oct 23. PMID 24152055
- See also: Division of Research, Department of Family & Community Medicine — http://dorfam.sw.org

RESULTS

PARTICIPANT FLOW:
Groups:
- CDSMP: 6-week educational classes
  CDSMP : 6-week classes
- Personal Digital Assistant (PDA): Personal digital assistance (technological)
  PDA : Technological assistance
- PDA/CDSMP: Combined intervention
  PDA/CDSMP : Combined technology and education
Period: Overall Study
Arm/Group | CDSMP | Personal Digital Assistant (PDA) | PDA/CDSMP | Control
Started | 101 | 81 | 99 | 95
Completed | 86 | 47 | 57 | 73
Not Completed | 15 | 34 | 42 | 22
Not completed — Non-Compliant or Unable to Contact | 15 | 12 | 15 | 20
Not completed — Withdrawal by Subject | 0 | 22 | 27 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDSMP | Personal Digital Assistant (PDA) | PDA/CDSMP | Control | Total
Number analyzed (Participants) | 101 | 81 | 99 | 95 | 376
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 81 | 56 | 73 | 70 | 280
  >=65 years | 20 | 25 | 26 | 25 | 96
Age Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.8) | 57.7 (10.8) | 57.7 (10.3) | 58.5 (11.9) | 57.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 47 | 53 | 53 | 207
  Male | 47 | 34 | 46 | 42 | 169
Region of Enrollment [Number; unit: participants]
  United States | 101 | 81 | 99 | 95 | 376
Minority [Number; unit: Participants] — Individuals categorized as minority were those who self-reported as either African American or Hispanic
  Participants
    No | 60 | 51 | 65 | 63 | 239
    Yes | 41 | 30 | 34 | 32 | 137
Race-Ethnicity [Number; unit: Participants]
  Non-Hispanic White | 58 | 49 | 61 | 58 | 226
  Non-Hispanic Black | 21 | 11 | 12 | 17 | 61
  Hispanic | 20 | 19 | 22 | 15 | 76
  Other | 2 | 2 | 4 | 5 | 13
Education [Number; unit: Participants]
  Less than high school | 6 | 4 | 3 | 3 | 16
  Some high school | 4 | 3 | 8 | 1 | 16
  High school graduate | 16 | 20 | 17 | 21 | 74
  Some college/vocational school | 46 | 34 | 33 | 36 | 149
  College graduate | 16 | 13 | 24 | 21 | 74
  Graduate school | 13 | 7 | 14 | 13 | 47
Income [Number; unit: Participants]
  < $15,000 | 12 | 11 | 7 | 9 | 39
  $15,000 - $24,999 | 11 | 14 | 19 | 16 | 60
  $25,000 - $49,999 | 41 | 37 | 32 | 30 | 140
  $50,000 - $75,000 | 12 | 12 | 23 | 17 | 64
  > $75,000 | 12 | 6 | 14 | 14 | 46
  Prefer not to answer | 13 | 1 | 4 | 9 | 27
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.5 (8) | 35.3 (7.3) | 34.6 (6.3) | 33.9 (7.7) | 34.3 (7.4)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm/Hg] | 131.9 (14.1) | 138.5 (21.2) | 136.2 (19.1) | 132.9 (21.7) | 134.8 (19.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm/Hg] | 79.4 (9.8) | 73.6 (11) | 78.8 (11.4) | 75.8 (13.6) | 77 (11.7)
HbA1c [Mean (Standard Deviation); unit: %] | 9.4 (1.7) | 9.3 (1.6) | 9.2 (1.4) | 9.2 (1.6) | 9.3 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Measures of HbA1c were collected from electronic health records dating back six months prior to orientation to the last day of study participation (45 days after the 12-month follow-up period). If a participant did not have any HbA1c value within the electronic health record for any particular follow-up visit, a lab test was scheduled to obtain a measure. Of the HbA1c collected six months prior to orientation, the value measured closest to the orientation date was considered as the baseline HbA1c value. HbA1c values that were measured on dates preceding the baseline HbA1c were not included; i.e., HbA1c values included in the analysis were those collected since the baseline HbA1c and until the last day of study participation.
Time Frame: 12 months
Population: A participant was included in the analysis if he/she had a HbA1c value collected. A longitudinal analysis was performed, with participants contributing one or more HbA1c values to the model. As such, all participants had at least one HbA1c value and were therefore included in the model.
Measure: Mean (Standard Deviation); unit: percentage of gycosylated HbA1c
Units Other Than Participants: HbA1c
Arm/Group | CDSMP | Personal Digital Assistant (PDA) | PDA/CDSMP | Control
Number analyzed (Participants) | 101 | 81 | 99 | 95
Number analyzed (HbA1c) | 388 | 267 | 307 | 365
percentage of gycosylated HbA1c | 8.7 (1.9) | 8.7 (1.7) | 8.6 (1.4) | 8.4 (1.6)
Statistical Analysis 1: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; We used a multilevel statistical model including time (in days) as a continuous variable, where 0=baseline. The lowest level of the hierarchy was repeated measurements of HbA1c on each subject, with participants themselves constituting the 2nd level. Forward selection was utilized, in which powers of time were added one at a time to the base model including treatment group effects. Interaction terms between time & treatment effects were added gradually and evaluated with likelihood ratio tests; Test type: Superiority or Other; p = 0.771, Likelihood Ratio Tests — A priori threshold for statistical significance is <0.05

2. Secondary Outcome: BMI
Description: Body mass index
Time Frame: 12 months
Population: BMI was computed from height & weight measurements from the 12-month follow-up (f/u) visit. Those unable to come in had height and weight abstracted from their EHRs. Measures recorded fell within the range of 10 days prior to and 45 days after participants' f/u visit dates. Those missing this information was not included in the analysis.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | CDSMP | Personal Digital Assistant (PDA) | PDA/CDSMP | Control
Number analyzed (Participants) | 67 | 30 | 39 | 56
kg/m^2 | 34.9 (9.2) | 35.8 (7.6) | 32.8 (5.5) | 33.9 (8.4)
Statistical Analysis 1: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; Test type: Superiority or Other; p = 0.2176, Regression, Linear — A priori threshold for statistical significance is <0.05; Robust variance estimates

3. Secondary Outcome: Patient Self-reported Perceived Health Status
Time Frame: 12 months
Population: Perceived health status was collected using a questionnaire administered during the 12-month follow-up visit. Individuals who did not complete the questionnaire during the follow-up visit or who refused to answer the question were not included in the analysis.
Measure: Number; unit: participants
Arm/Group | CDSMP | Personal Digital Assistant (PDA) | PDA/CDSMP | Control
Number analyzed (Participants) | 46 | 11 | 20 | 30
participants
  Excellent | 3 | 0 | 1 | 1
  Very Good | 13 | 3 | 6 | 5
  Good | 19 | 6 | 4 | 14
  Fair | 10 | 2 | 9 | 8
  Poor | 1 | 0 | 0 | 2
Statistical Analysis 1: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; Test type: Superiority or Other; p = 0.572, Fisher Exact — A priori threshold for statistical significance was <0.05

4. Secondary Outcome: Diabetes-related Behaviors
Description: Participants were asked the number of days in the past 7 which they participated in various diabetes self-care activities on diet, exercise, home blood glucose monitoring, and foot care.
Time Frame: 12 months
Population: Those who completed a questionnaire at baseline and at their 12-month visit were included. Also, they had to have answered questions regarding self-care activities on both surveys since the calculated mean was the average difference in days within the past 7 that individuals participated in self-care activities between 12-months and baseline.
Measure: Mean (Standard Deviation); unit: Days (e.g., Avg diff 12mo vs baseline)
Arm/Group | CDSMP | Personal Digital Assistant (PDA) | PDA/CDSMP | Control
Number analyzed (Participants) | 46 | 11 | 20 | 30
Days (e.g., Avg diff 12mo vs baseline)
  Test blood sugar | 0.26 (3.01) | -0.91 (2.12) | 0.10 (2.05) | 0.97 (2.76)
  Test blood sugar the recommended times | 0.55 (3.37) | -1.22 (2.28) | 0.11 (2.40) | 1.21 (3.28)
  Exercise at least 30 minutes | 0.80 (2.90) | 0.09 (2.39) | -0.16 (2.22) | 0.70 (2.44)
  Participate in a specific exercise session | 0 (2.39) | -1.00 (1.61) | 0.37 (1.89) | 0.72 (3.06)
  Check feet | 1.84 (2.99) | 0.36 (2.11) | 0.65 (2.66) | 0.63 (3.11)
  Wash feet | 0.52 (1.55) | 0.09 (1.70) | -0.05 (1.00) | -0.17 (1.37)
  Soak feet | 0.74 (2.29) | 1.00 (2.00) | 0.55 (2.50) | 0.32 (3.13)
  Dry between toes | 0.53 (2.52) | 0.36 (1.91) | 1.53 (3.04) | 0.76 (2.67)
  Inspect inside of shoes | 1.47 (3.53) | 0.82 (1.89) | 0.20 (3.16) | 0.11 (3.57)
  Follow healthful eating plan | 0.28 (2.05) | -0.36 (1.96) | 0.60 (2.44) | 0.93 (2.45)
  Space carbohydrates | 0.15 (3.00) | -0.36 (3.67) | 0.60 (2.58) | 0.64 (2.28)
  Eat 5+ servings of fruits and vegetables | 0.31 (2.92) | 0.64 (2.46) | 0.35 (2.06) | 1.10 (2.14)
  Eat high-fat foods | -0.98 (2.17) | 1.45 (2.34) | 0.53 (2.29) | -0.72 (2.20)
  Eat packaged foods (e.g., sweets and desserts) | -0.09 (2.26) | 0 (0.63) | 0 (2.68) | -0.66 (2.02)
  Followed a healthful eating plan | 0.32 (1.97) | -0.36 (1.63) | 0.50 (2.37) | 0.52 (2.34)
Statistical Analysis 1: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Test blood sugar."; Test type: Superiority or Other; p = 0.26, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Test blood sugar the recommended times."; Test type: Superiority or Other; p = 0.21, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Exercise at least 30 minutes."; Test type: Superiority or Other; p = 0.53, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Participate in a specific exercise session."; Test type: Superiority or Other; p = 0.24, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Check feet."; Test type: Superiority or Other; p = 0.18, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Wash feet."; Test type: Superiority or Other; p = 0.19, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 7: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Soak feet."; Test type: Superiority or Other; p = 0.87, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 8: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Dry between toes."; Test type: Superiority or Other; p = 0.53, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 9: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Inspect inside of shoes."; Test type: Superiority or Other; p = 0.32, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 10: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Follow healthful eating plan."; Test type: Superiority or Other; p = 0.37, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 11: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Space carbohydrates."; Test type: Superiority or Other; p = 0.72, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 12: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Eat 5+ servings of fruits and vegetables."; Test type: Superiority or Other; p = 0.59, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 13: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Eat high-fat foods."; Test type: Superiority or Other; p < 0.004, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 14: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Eat packaged foods (e.g., sweets and desserts)."; Test type: Superiority or Other; p = 0.66, ANOVA — A priori threshold for statistical significance is <0.05
Statistical Analysis 15: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the average difference in days for the diabetes self-care activity, "Followed a healthful eating plan."; Test type: Superiority or Other; p = 0.68, ANOVA — A priori threshold for statistical significance is <0.05

5. Secondary Outcome: Quality of Life (QOL)
Description: Participants where asked the number of days in the past 30 days in which their physical (phys) and/or mental was not good, and whether their usual activity was affected by their physical/mental health.
Time Frame: 12 months
Population: Participants were included if they completed the 12-mo follow-up questionnaire. They also had to have answered questions pertaining to quality of life. Missing responses were not included.
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | CDSMP | Personal Digital Assistant (PDA) | PDA/CDSMP | Control
Number analyzed (Participants) | 46 | 11 | 20 | 30
Number of days
  Physical health was not good in the past 30 days | 5.9 (8.7) | 9.0 (11.7) | 8.5 (10.2) | 7.3 (8.8)
  Mental health was not good in the past 30 days | 6.8 (9.6) | 7.2 (12.6) | 7.3 (11.0) | 6.6 (10.2)
  Poor phys/mental health prevented usual activities | 3.8 (7.2) | 7.3 (12.6) | 7.8 (9.1) | 5.4 (9.3)
Statistical Analysis 1: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the quality of life measure, "Number of days physical health was not good in the past 30 days" at the 12 month follow-up visit; Test type: Superiority or Other; p = 0.685, Regression, Linear — A priori threshold for statistical significance is <0.05; Robust Variance Estimation
Statistical Analysis 2: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the quality of life measure, "Number of days mental health was not good in the past 30 days" at the 12 month follow-up visit; Test type: Superiority or Other; p = 0.997, Regression, Linear — A priori threshold for statistical significance is <0.05; Robust variance estimation
Statistical Analysis 3: Comparison: CDSMP vs Personal Digital Assistant (PDA) vs PDA/CDSMP vs Control; This analysis was to compare the quality of life measure, "Number of days poor physical/mental health prevented usual activity in the past 30 days" at the 12 month follow-up visit; Test type: Superiority or Other; p = 0.3067, Regression, Linear — A priori threshold for statistical significance is <0.05; Robust variance estimation

ADVERSE EVENTS:
Arm/Group | CDSMP | Personal Digital Assistant (PDA) | PDA/CDSMP | Control
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/81 | 0/99 | 0/95
Other Adverse Events (participants affected / at risk) | 0/101 | 0/81 | 0/99 | 0/95

LIMITATIONS AND CAVEATS:
Differential dropout across interventions. Failure to obtain 50% minority and 50% non-minority participants, preventing further analyses regarding race/ethnicity differences in outcome. Could only provide information in an exploratory manner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No